CLINICAL TRIAL: NCT07174024
Title: A Comparative Study on the Efficacy of Blue Light Emitting Diodes Therapy Versus Targeted Narrow Band UVB in Stable Non-segmental Vitiligo Patients.
Acronym: Nb-UVB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Maher Mahmoud Mahran, Lecturer of Dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-92-2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Vitiligo
Keywords: blue light emitting diode
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients will receive NB-UVB phototherapy sessions on a Randomly selected patch (Active Comparator): patients will receive NB-UVB phototherapy sessions on a Randomly selected patch
  Interventions: Device: Narrow Band UVB Treatment
- Patients will receive blue light emitting diodes phototherapy on a randomly selected patch (Active Comparator): Patients will receive blue light emitting diodes phototherapy on a randomly selected patch
  Interventions: Device: blue light emitting diode

INTERVENTIONS:
Device: Narrow Band UVB Treatment — type of phototherapy
  Arms: patients will receive NB-UVB phototherapy sessions on a Randomly selected patch
Device: blue light emitting diode — type of diode
  Arms: Patients will receive blue light emitting diodes phototherapy on a randomly selected patch

SUMMARY:
A comparative study on the efficacy of blue light emitting diodes therapy versus targeted Narrow band UVB in stable non-segmental vitiligo patients.

DETAILED DESCRIPTION:
A comparative study on the efficacy of blue light emitting diodes therapy versus targeted Narrow band UVB in stable non-segmental vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* All age group.

  * Both genders.
  * Subjects with stable non-segmental vitiligo (≥2 patches) acral or non-acral patches of diameter ≤ 2cm.

Exclusion Criteria:

* Prior treatment with laser therapies for at least 3 months

  * Recent exfoliation procedures.
  * Recent surgical procedures.
  * Poor skin conditions including keloids.
  * Hypersensitivity to light ( visible and near-infrared).
  * Medications that make users more sensitive to light.
  * Anticoagulant and immunosuppressive treatments.
  * Gestations or breastfeeding.
  * A personal or family history of skin cancer.
  * Unstable vitiligo (older lesions have not progressed for the last 1 years and lack of Koebner phenomena ).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-23 (Actual)

PRIMARY OUTCOMES:
Assess the degree of improvement in vitiligo pigmentation using VASI scores before and after treatment. | 48 weeks
  Assess the degree of improvement in vitiligo pigmentation using VASI scores before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No